CLINICAL TRIAL: NCT05265104
Title: Clinical and Radiographic Evaluation of the Efficacy of Laser Versus Silver Diamine Flouride (SDF) in Hall Technique in Primary Teeth
Brief Title: Laser Versus Silver Diamine Fluoride in Hall Technique in Primary Teeth
Acronym: SDF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Rasha Farouk Sharaf, Researcher of Pediatric Dentistry, National Research Centre, Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1434052021
Record Dates: First submitted 2022-02-03; First posted 2022-03-03 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Carious Teeth
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SDF with stainless steel crown (Experimental): mixture of silver , diamine and fluoride applied using a brush to the caries in the primary molar , it is used to arrest the progress of the carious lesion
  Interventions: Drug: SDF with stainless steel crown
- Diode laser with stainless steel crown (Experimental): Diode laser beam is used to sterilize the carious lesions to arrest the progress of the dental caries
  Interventions: Device: Diode laser application with stainless steel crown
- Control, stainless steel crown only (Active Comparator): stainless steel crown is cemented on the carious primary molar to arrest the progress of the caries, by isolating the tooth from the surrounding bacteria, this is the concept of the Hall technique.
  Interventions: Other: stainless steel crown only

INTERVENTIONS:
Drug: SDF with stainless steel crown — Silver Diamine Fluoride (38%) applied to the carious lesion in the primary molars with a brush and the tooth is sealed with a stainless steel crown
  Arms: SDF with stainless steel crown
Device: Diode laser application with stainless steel crown — Diode laser will be applied to the carious lesions primary molars to eradicate the bacteria and then the tooth will be sealed with stainless steel crown
  Arms: Diode laser with stainless steel crown
Other: stainless steel crown only — the primary molars with carious lesions will be sealed with stainless steel crowns following the concept of hall technique
  Arms: Control, stainless steel crown only

SUMMARY:
The hall technique for primary teeth depends on the idea of isolation of the carious non exposed primary tooth from all bacteria present in the oral cavity by using a stainless-steel crown which result in arresting of the caries and preventing its progress to the pulp. Recently laser and Silver Diamide Fluoride (SDF) have been used to arrest the progress of caries so in the current study we will compare the success rate of hall technique with either laser or SDF in arresting of caries

DETAILED DESCRIPTION:
The high frequency of caries in primary teeth and its inadequate treatment are major public health problems during childhood. Nowadays, the Hall technique is one of the methods used for biological sealing in carious lesions in primary molars. Thus, the bacteria will be sealed from oral environment and the caries will be inactive. Using the Hall technique, the crown is placed without local anesthesia, caries removal, or tooth preparation. Then, the crown is fitted over the carious primary molar by either the dentist's finger pressure, or the child's biting force. The average results of many clinical trials showed that the success rates of the Hall technique were greater than the conventional restorations. However, some criteria of minor failures were seen in 26.6% of Hall crowns. Silver diamine fluoride (SDF), a clear liquid that combines the antibacterial effects of silver and the remineralizing effects of fluoride, is a promising therapeutic agent for managing caries lesions in young children, its effectiveness in reducing specific cariogenic bacteria and its remineralizing potential on enamel and dentin have been reported in many studies. Recently, lasers have been proven to significantly arrest the dental caries by increasing the acid resistance of the enamel with an antibacterial effect. Diode lasers with several positive aspects, such as the small size, low cost, and ease of use in the oral cavity, were found to have a caries prevention and arrest effect on the dental enamel, particularly deciduous teeth. In the current study the success rate of Hall technique using SDF will be compared to the same technique using Diode laser in arresting the carious lesions in primary teeth.

ELIGIBILITY:
Inclusion Criteria:

* Patients should be medically free
* Presence of asymptomatic enamel and dentin caries in one or more primary molars, which can be detected clinically and radiographically
* Periapical radiograph should show caries involving the outer half of the dentin
* There should be no signs or symptoms of pulpal pathosis

Exclusion Criteria:

* Immunocompromised patients
* Presence of any signs or symptoms of pulpal pathosis denoting irreversible pulpitis
* Parents who are not willing to come in the follow up visits

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Pain on biting | 1 year
  Verbal questioning of the patient
gingival swelling | 1 year
  visual examination by the operator

SECONDARY OUTCOMES:
Periapical/ furcation radiolucency | 1 year
  perapical radiograph using paralleling technique by DE GOTZEN XGENUS intra-oral x ray unit

CONTACTS AND LOCATIONS:
Overall Officials: Rasha Sharaf, PhD, Principal Investigator — Researcher at the National Research Centre
Locations (1):
- Dr. Rasha Farouk Sharaf, Cairo, Egypt

REFERENCES:
- [Background] Chaurasiya A, Gojanur S. Evaluation of the clinical efficacy of 38% silver diamine fluoride in arresting dental caries in primary teeth and its parental acceptance. J Indian Soc Pedod Prev Dent. 2021 Jan-Mar;39(1):85-89. doi: 10.4103/jisppd.jisppd_34_21. PMID 33885393
- [Result] Altoukhi DH, El-Housseiny AA. Hall Technique for Carious Primary Molars: A Review of the Literature. Dent J (Basel). 2020 Jan 17;8(1):11. doi: 10.3390/dj8010011. PMID 31963463
- [Result] Clark W, Geneser M, Owais A, Kanellis M, Qian F. Success rates of Hall technique crowns in primary molars: a retrospective pilot study. Gen Dent. 2017 Sep-Oct;65(5):32-35. PMID 28862586
- [Result] Crystal YO, Niederman R. Evidence-Based Dentistry Update on Silver Diamine Fluoride. Dent Clin North Am. 2019 Jan;63(1):45-68. doi: 10.1016/j.cden.2018.08.011. PMID 30447792
- [Result] Chokhachi Zadeh Moghadam N, Seraj B, Chiniforush N, Ghadimi S. Effects of Laser and Fluoride on the Prevention of Enamel Demineralization: An In Vitro Study. J Lasers Med Sci. 2018 Summer;9(3):177-182. doi: 10.15171/jlms.2018.32. Epub 2018 Jul 28. PMID 30809328